CLINICAL TRIAL: NCT07093151
Title: COMparison of Postcraniotomy Blood pressurE Target Effectiveness (COMPETE)
Brief Title: Comparison of Post-Craniotomy Blood Pressure Targets
Acronym: COMPETE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Patrick Kelly, Principal Investigator, Assistant Professor of Neurological Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 250498
Record Dates: First submitted 2025-07-19; First posted 2025-07-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Hemorrhage, Hypertensive; Craniotomy Tumor Removal Surgery
Keywords: Perioperative Care; Post-Craniotomy Emergence Hypertension
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator Arm 1: SBP target <160 mmHg (Active Comparator): The neuro-intensive care team will monitor the patient's SBP and treat with antihypertensive medications to achieve an SBP<160mHg. Selection of the appropriate oral or IV medication is at the discretion of the neuro-ICU team; most frequently used agents clinically include nicardipine, labetalol, and hydralazine. Selection of the appropriate agent is based on other clinical elements including severity of hypertension, heart rate, patients' home medication regimens, and any medication interactions or allergies. The blood pressure goal will be continued throughout the hospitalization. The arterial line will be removed at the discretion of the neurosurgery team, typically on the morning of the first day after surgery.
  Interventions: Other: Target SBP <160mmHg
- Comparator Arm 2: SBP Target <140 mmHg (Active Comparator): The neuro-intensive care team will monitor the patient's SBP and treat with antihypertensive medications to achieve an SBP<140mHg. Selection of the appropriate oral or IV medication is at the discretion of the neuro-ICU team, as described above for Comparator Arm 1. The blood pressure goal will be maintained until the neurosurgery team chooses to 'liberalize' the blood pressure goal to higher SBP levels. The arterial line will be removed when the blood pressure goal is liberalized, typically on the morning of the first day after surgery.
  Interventions: Other: Target SBP <140 mmHg

INTERVENTIONS:
Other: Target SBP <160mmHg — For subjects assigned to the SBP <160 mmHg group, an SBP target order will be placed to guide the neuro-intensive care team to treat the patient with antihypertensive medications as needed to achieve an SBP <160 mmHg. Selection of the antihypertensive medication and administration route is at the discretion of the treating team. Patients will undergo regular and frequent blood pressure measurements using the arterial line placed during surgery, or through a non-invasive blood pressure measurement method if no arterial line is present.
  Arms: Comparator Arm 1: SBP target <160 mmHg
Other: Target SBP <140 mmHg — For subjects assigned to the SBP <140 mmHg group, an SBP target order will be placed to guide the neuro-intensive care team to treat the patient with antihypertensive medications as needed to achieve an SBP <140 mmHg. Selection of the antihypertensive medication and administration route is at the discretion of the treating team. Patients will undergo regular and frequent blood pressure measurements using the arterial line placed during surgery, or through a non-invasive blood pressure measurement method if no arterial line is present.
  Arms: Comparator Arm 2: SBP Target <140 mmHg

SUMMARY:
The goal of this pragmatic clinical trial is to learn if a more intensive or more liberal blood pressure target after surgery is more effective in improving patient outcomes for adults undergoing craniotomy for removal of a brain tumor. There is little evidence to help doctors decide the best post-operative blood pressure target for their patients. The main question this study aims to answer is if patients with a post-operative systolic blood pressure target of <160 mmHg will have a shorter hospital length of stay than those with a blood pressure target of <140 mmHg, without increasing the rate of post-operative bleeding in the brain.

DETAILED DESCRIPTION:
Over 160,000 craniotomies, a type of brain surgery, are performed annually in the United States. High blood pressure is believed to increase the risk of post-operative bleeding in the brain, known as intracranial hemorrhage (ICH). This perceived risk has led many doctors to impose post-operative systolic blood pressure (SBP) limits, with aggressive treatment when SBP rises above the target thresholds. The use of intensive SBP goals often requires antihypertensive medication treatment, occasionally including intravenous (IV) drips. These medical therapies could have several adverse effects related to end-organ function. Additionally, close SBP monitoring with an arterial line and/or treatment with IV antihypertensives often requires intensive care unit (ICU) level of care. 40% of academic medical programs use a goal of SBP<160mmHg as supported by this limited evidence, while 45% of programs use an even more stringent SBP goal of <140mmHg.

This study is a single-center, pragmatic, randomized trial comparing the effectiveness of these two standard-of-care post-craniotomy SBP goals in reducing patient hospital length of stay, risk of ICH, and adverse side effects of antihypertensive use. Eligible patients will be randomized to receive an order for a target SBP <140 mmHg or SBP <160 mmHg during this period. We hypothesize that a target SBP <160 mmHg will decrease patient hospital length of stay without increasing the risk of ICH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Undergoes craniotomy for resection of an intradural brain tumor scheduled using any of the following Current Procedural Terminology (CPT) codes: 61304, 61305, 61330, 61333, 61510, 61512, 61516, 61518, 61519, 61520, 61521, 61524, 61526, 61530, 61545, 61580, 61581, 61582, 61583, 61584, 61585, 61586, 61590, 61591, 61592, 61595, 61596, 61597, 61598, 61600, 61601, 61605, 61606, 61607, 61608, 61615, 61616

Exclusion Criteria:

* Declines to consent
* Attending decisions based on intraoperative findings (i.e. attending physician does not have equipoise that either blood pressure threshold would be acceptable for the post-operative care of the patient).
* Patient is a prisoner
* Patient is known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | From enrollment to first hospital discharge or 90 days, whichever is sooner
  Length of patient hospital stay in days

SECONDARY OUTCOMES:
ICU length of stay | From enrollment to transfer out of the ICU or 90 days, whichever is sooner.
  Length of patient stay in the Neuro Intensive Care Unit after craniotomy
Intracranial hemorrhage (ICH) incidence | From enrollment to hospital discharge
  Rate of intracranial hemorrhage requiring return to the operating room
Patient-Reported Outcome Measurement Information System-10 (PROMIS10) score | From enrollment to 90 days following enrollment
  PROMIS10 responses collected at routine postoperative neurosurgery clinic follow-up visits. The PROMIS Global 10 uses T-scores to interpret results. T-scores are standardized scores with a mean of 50 and a standard deviation of 10.
Functional Assessment of Cancer Therapy - Brain (FACT-Br) score | From enrollment to 90 days following enrollment.
  FACT-Br responses collected at routine postoperative neurosurgery clinic follow-up visits. This scale is measured on a 5 point Likert-type scale, with higher scores indicating better quality of life.
Composite of adverse end-organ hypoperfusion events related to antihypertensive use | From enrollment to hospital discharge or 90 days, whichever is sooner.
  Composite measure of inpatient mortality, acute kidney injury, BNP elevation, and myocardial infarction during hospital stay.

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made accessible to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.